CLINICAL TRIAL: NCT06925282
Title: Determinants of Rescue Ventilation Requirement in Airway Surgery Under General Anesthesia With Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): A Prospective Observational Study
Brief Title: Determinants of Rescue Ventilation Requirement in Airway Surgery Under General Anesthesia With THRIVE
Acronym: THRIVE
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Shin Kyung Won, MD, Clinical instructor, Seoul National University Hospital
Other Study IDs: 2503-107-1622
Record Dates: First submitted 2025-03-31; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Subglottic Stenosis (SGS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- THRIVE: Adult patients undergoing airway surgery under general anesthesia with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE).

SUMMARY:
The anesthesia and surgical procedures from the time the patient enters the operating room to discharge from the recovery room are identical to those used in conventional airway surgeries performed under general anesthesia with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE). The time point at which rescue ventilation is required due to a drop in oxygen saturation below 92% during anesthesia will be recorded, and the predictive factors for this event will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective airway surgery under general anesthesia with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE)
* Patients who provide written informed consent

Exclusion Criteria:

* Patients who decline to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled to undergo elective airway surgery under general anesthesia with THRIVE at a single tertiary academic hospital. A total of 80 patients will be prospectively enrolled. All participants will receive standard anesthetic care, and data will be collected during the intraoperative period for analysis of factors associated with the requirement for rescue ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Time to Rescue Ventilation Due to Hypoxemia During Airway Surgery With THRIVE Under General Anesthesia | From the start of apnea to the initiation of rescue ventilation during surgery (intraoperative period)
  The primary outcome is the time from the start of apnea to the initiation of rescue ventilation, defined as the point when oxygen saturation (SpO₂) falls to 92% or below during airway surgery under general anesthesia with Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE). This will be measured using continuously recorded intraoperative data. The aim is to identify clinical predictors (e.g., anatomical and physiological variables) associated with the need for rescue ventilation.

SECONDARY OUTCOMES:
Lowest Oxygen Saturation After Initiation of Rescue Ventilation | From the start of apnea to the initiation of rescue ventilation during surgery (intraoperative period)
  This outcome measures the lowest oxygen saturation (SpO₂) observed after the initiation of rescue ventilation during airway surgery with THRIVE under general anesthesia. Data will be extracted from intraoperative monitoring records.
Time to Recovery of SpO₂ to 100% After Rescue Ventilation | From the start of apnea to the initiation of rescue ventilation during surgery (intraoperative period)
  This outcome measures the time interval from the start of rescue ventilation to the recovery of oxygen saturation (SpO₂) to 100%. The measurement will help evaluate the efficacy of rescue ventilation in restoring oxygenation.
End-Tidal CO₂ at the Time of Rescue Ventilation | From the start of apnea to the initiation of rescue ventilation during surgery (intraoperative period)
  This outcome records the end-tidal carbon dioxide (EtCO₂) level at the moment rescue ventilation is initiated. It aims to assess the extent of CO₂ retention during apnea and its relationship to the timing of rescue ventilation.
Predictive Factors for the Requirement of Rescue Ventilation | From the start of apnea to the initiation of rescue ventilation during surgery (intraoperative period)
  This outcome involves analysis of patient anatomical and physiological factors (e.g., Mallampati class, thyromental distance, neck circumference, presence of retrognathia) to determine their association with the need for rescue ventilation during THRIVE-supported airway surgery.